CLINICAL TRIAL: NCT02495714
Title: HOPPLearning - Active Learning in Elementary Schools in Horten Municipality
Brief Title: HOPPLearning - Active Learning in Elementary Schools
Acronym: HOPPLearning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kristiania University College (Other)
Collaborators: Horten municipality (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KristianiaUC
Record Dates: First submitted 2015-06-20; First posted 2015-07-13 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Health Behaviour
Keywords: Exercise; Diet; Learning
MeSH Terms: conditions — Motor Activity | interventions — Supervised Machine Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention schools (Experimental): Active Learning; One hour each schoolday of physical Activity as part of academic learning Dietary councelling; teaching children and parents about a healty diet
  Interventions: Behavioral: Active learning; Behavioral: Dietary councelling
- Control schools (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Active learning — Physical activity one hour a day as part of academic learning
  Arms: Intervention schools
Behavioral: Dietary councelling — Teaching children and parents about a healthy diet
  Arms: Intervention schools

SUMMARY:
HOPP Learning will be implemented in elementary schools in the Horten municipality and will assess the effect of a combined pedagogical approach, active learning, on a large student population. Students are to increase their amount of physical activity with learning, during a school day by one hour.

DETAILED DESCRIPTION:
Background It has for many decades been a discussion whether the proportion of hours of physical activity should be increased in the Norwegian primary school. In light of the evolution of inactivity, overweight and obesity, both internationally and in Norway, it is now time to implement measures that can provide improved health and preventing lifestyle diseases among children and adolescents. Until now, one in Norwegian society based on the fact that children are active enough in their spare time, with sport as an arena. This assertion has had its validity, but not with the tendency of children are significantly more sedentary than their parents were in their infancy. Thus, the community must take more responsibility. One of the measures is to increase the physical activities offered in primary schools. Then all the children get the opportunity to form healthy habits with regular physical activity.

HOPP Learning will be implemented in elementary schools in the Horten municipality and will assess the effect of a combined pedagogical approach, active learning, on a large student population. Students are to increase their amount of physical activity, during a school day by one hour. To evaluate the effect of HOPP Learning Horten municipality contacted University College of Health Sciences - Campus Kristiania.

Aims The primary aim is to chart and assess the effect of active learning through analysis of dietary intake (Ungkost 2000 questionnaire), quality of life (ILC questionnaire), cognitive tests (computer based measurements of reaction time using Flanker and Stroop test), academic performance (grades in national tests) and physiological factors as activity level (accelerometer measurements), aerobic capacity (Andersen shuttle run test and oxygen uptake), balance (Balance Y-test) and strength (Jamar handgrip). In addition medical variables as blood pressure, peak expiratory flow and blood work (total cholesterol, HDL, iron, feritin, CRP, blood sugar, Hb, Hematocrit, RBC).

Sample The project has a prospective clinical controlled study design and involves seven elementary schools in Horten Municipality with the estimated number of children in 1-6 grade being 1,822. The 12 year olds in the current schools will not be tested when they go over to their respective secondary schools in 2016 so will not participate in the intervention. Similarly, those children who start 1st grade in 2015 not be included in the intervention as they are enrolled in kindergarten during the first round of tests in Spring 2015. Consequently there will be a calculated "drop off" of one school grade per year based on the selection from the initial testing during spring 2015, and from the second round of testing in 2016. Based on an analysis of socioeconomic status between municipalities in Norway, Loerenskog and Baerum municipality has a socioeconomic composition as Horten. Given health inequalities in children are directly related to parents' socioeconomic status, and in particular education, Loerenskog and Baerum municipality were chosen as the control population. Two elementary schools were contacted and agreed to participate as control schools, ca. 500 pupils at each school. Similarly calculated dropout rates will occur at the control school. The total inclusion sample is approximately 2,800 pupils. Inclusion criteria: Students from Grade 1-6 from all elementary schools in Horten municipality and from two control schools. Exclusion criteria: Students with psychological or physical disabilities that prevent them participating in the tests, students afflicted with sickness/disease during the testing period and students who do not wish to participate in the test.

Implementation of the intervention A large activity learning library within reading, mathematics and english within the academic guidelines for grades 1-7 has been established. There is thus a total of 32 sites where it is 510 activities within each step. This means that it is unique exercise sets distributed on grades and subjects the individual teachers will have at least one hour per class they are responsible for every day. The range of exercises are based both on the teachers' own ideas, proposals from the Education directorate and www.skolesekken.no. Horten Municipality has distributed this exercise library to the individual schools. The activity is organized as different activity programs of 15 minutes for each subject they wish to teach.

Combining physical activity and learning (basic subjects) exercise sets are stored in boxes with the accompanying learning tools: a crate for english 1st grade, a crate for English 2nd grade, etc., thus making it easy to begin a lesson by simply bringing a box to each class.

ELIGIBILITY:
Inclusion Criteria:

* Students from Grade 1-6 (2015) from all elementary schools in Horten municipality and two schools from Loerenskog and Baerum municipality.

Exclusion Criteria:

* Students with psychological and physical disabilities preventing them participating in the tests
* Students afflicted with sickness/disease during the testing period
* Students who do not wish to participate in the test

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2300 (Actual)
Dates: Start 2015-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Academic performance | 72 months
  Change in academic performance due to change in the pedagogic technique using standarised national academic tests

SECONDARY OUTCOMES:
Cognitive ability | 72 months
  Measurements of cognitive ability pre- and post intervention using Eriksen Flanker test and Stroop test
Diet changes | 72 months
  Based on diet information to the parents diet change in the children are measured using a questionnaire Ungkost 2000
Changes in quality of life | 72 months
  The intervention may change QOL. The study is using ILC for parents and children to measure the change
Changes in blood values | 72 months
  Blood values of total cholesterol, HDL, 6-months blood-sugar, Hb, RBC, Haematocrit, ferritin, iron and CRP are measured pre- and post intervention.
General physical capacity | 72 months
  General physical capacity is measured in all participants using Andersen shuttle run test, Jamar handgrip, Balance Y-test and maximal oxygen uptake (1st. grade). Changes are expected due to increased physical activity level.
Cardiovascular risk factors | 72 months
  The change in cardiovascular risk factors during 5 years of intervention is measured using a combination of data from medical tests, physiological tests and questionnaires
Physical activity level | 12 months
  Change in physical activity level due to active learning are measured using Actigraph wGT3X-BT across one week

CONTACTS AND LOCATIONS:
Overall Officials: Per Morten Fredriksen, Professor, Principal Investigator — University College of Health Sciences - Campus Kristiania
Locations (1):
- Kristiania University College, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Onis M, Blossner M, Borghi E. Global prevalence and trends of overweight and obesity among preschool children. Am J Clin Nutr. 2010 Nov;92(5):1257-64. doi: 10.3945/ajcn.2010.29786. Epub 2010 Sep 22. PMID 20861173
- [Background] Wedderkopp N, Froberg K, Hansen HS, Andersen LB. Secular trends in physical fitness and obesity in Danish 9-year-old girls and boys: Odense School Child Study and Danish substudy of the European Youth Heart Study. Scand J Med Sci Sports. 2004 Jun;14(3):150-5. doi: 10.1111/j.1600-0838.2004.00365.x. PMID 15144354
- [Background] Moller NC, Wedderkopp N, Kristensen PL, Andersen LB, Froberg K. Secular trends in cardiorespiratory fitness and body mass index in Danish children: The European Youth Heart Study. Scand J Med Sci Sports. 2007 Aug;17(4):331-9. doi: 10.1111/j.1600-0838.2006.00583.x. Epub 2006 Aug 10. PMID 16903897
- [Background] Tomkinson GR, Olds TS. Secular changes in pediatric aerobic fitness test performance: the global picture. Med Sport Sci. 2007;50:46-66. doi: 10.1159/000101075. PMID 17387251
- [Background] Ekelund U, Anderssen SA, Froberg K, Sardinha LB, Andersen LB, Brage S; European Youth Heart Study Group. Independent associations of physical activity and cardiorespiratory fitness with metabolic risk factors in children: the European youth heart study. Diabetologia. 2007 Sep;50(9):1832-1840. doi: 10.1007/s00125-007-0762-5. Epub 2007 Jul 20. PMID 17641870
- [Background] Resaland GK, Mamen A, Anderssen SA, Andersen LB. Cardiorespiratory fitness and body mass index values in 9-year-old rural Norwegian children. Acta Paediatr. 2009 Apr;98(4):687-92. doi: 10.1111/j.1651-2227.2008.01181.x. Epub 2009 Jan 5. PMID 19133872
- [Background] Resaland GK, Mamen A, Boreham C, Anderssen SA, Andersen LB. Cardiovascular risk factor clustering and its association with fitness in nine-year-old rural Norwegian children. Scand J Med Sci Sports. 2010 Feb;20(1):e112-20. doi: 10.1111/j.1600-0838.2009.00921.x. Epub 2009 Jun 9. PMID 19522748
- [Background] Resaland GK, Andersen LB, Mamen A, Anderssen SA. Effects of a 2-year school-based daily physical activity intervention on cardiorespiratory fitness: the Sogndal school-intervention study. Scand J Med Sci Sports. 2011 Apr;21(2):302-9. doi: 10.1111/j.1600-0838.2009.01028.x. PMID 19895384
- [Background] Bugge A, Tarp J, Ostergaard L, Domazet SL, Andersen LB, Froberg K. LCoMotion - Learning, Cognition and Motion; a multicomponent cluster randomized school-based intervention aimed at increasing learning and cognition - rationale, design and methods. BMC Public Health. 2014 Sep 18;14:967. doi: 10.1186/1471-2458-14-967. PMID 25236478
- [Background] Fedewa AL, Ahn S. The effects of physical activity and physical fitness on children's achievement and cognitive outcomes: a meta-analysis. Res Q Exerc Sport. 2011 Sep;82(3):521-35. doi: 10.1080/02701367.2011.10599785. PMID 21957711
- [Background] Tomporowski PD, Davis CL, Miller PH, Naglieri JA. Exercise and Children's Intelligence, Cognition, and Academic Achievement. Educ Psychol Rev. 2008 Jun 1;20(2):111-131. doi: 10.1007/s10648-007-9057-0. PMID 19777141
- [Background] Singh A, Uijtdewilligen L, Twisk JW, van Mechelen W, Chinapaw MJ. Physical activity and performance at school: a systematic review of the literature including a methodological quality assessment. Arch Pediatr Adolesc Med. 2012 Jan;166(1):49-55. doi: 10.1001/archpediatrics.2011.716. PMID 22213750
- [Background] Brown T, Summerbell C. Systematic review of school-based interventions that focus on changing dietary intake and physical activity levels to prevent childhood obesity: an update to the obesity guidance produced by the National Institute for Health and Clinical Excellence. Obes Rev. 2009 Jan;10(1):110-41. doi: 10.1111/j.1467-789X.2008.00515.x. Epub 2008 Jul 30. PMID 18673306
- [Background] van Sluijs EM, McMinn AM, Griffin SJ. Effectiveness of interventions to promote physical activity in children and adolescents: systematic review of controlled trials. Br J Sports Med. 2008 Aug;42(8):653-7. PMID 18685076
- [Background] Kriemler S, Meyer U, Martin E, van Sluijs EM, Andersen LB, Martin BW. Effect of school-based interventions on physical activity and fitness in children and adolescents: a review of reviews and systematic update. Br J Sports Med. 2011 Sep;45(11):923-30. doi: 10.1136/bjsports-2011-090186. PMID 21836176
- [Derived] Fredriksen PM, Mamen A, Goswami N, Lindberg M. Waist-to-Height Ratio as a predictor of cardiovascular and metabolic health in a pediatric population. PLoS One. 2025 Jul 9;20(7):e0326772. doi: 10.1371/journal.pone.0326772. eCollection 2025. PMID 40632711
- [Derived] Fredriksen PM, Hjelle OP, Mamen A, Meza TJ, Westerberg AC. The health Oriented pedagogical project (HOPP) - a controlled longitudinal school-based physical activity intervention program. BMC Public Health. 2017 Apr 28;17(1):370. doi: 10.1186/s12889-017-4282-z. PMID 28454531